CLINICAL TRIAL: NCT05302648
Title: A Early Phase 1 Clinical Trial to Evaluate the Safety and Efficacy of Human Derived Anti-BCMA CAR-T Injection for Subjects with Relapsed/Refractory Multiple Myeloma
Brief Title: To Evaluate the Safety and Efficacy of Human Derived Anti-BCMA CAR-T Injection for Subjects with R/R MM
Status: Active, not recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Shanghai Changzheng Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN01-MM03-POC
Record Dates: First submitted 2022-03-03; First posted 2022-03-31 (Actual); Last update posted 2025-01-03 (Actual); Status verified 2024-12

CONDITIONS: Multiple Myeloma
Keywords: BCMA; CAR-T; multiple myeloma; Relapsed /Refractory
MeSH Terms: conditions — Multiple Myeloma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Human Derived anti-BCMA CAR-T Injection (Experimental): Single administration：1.0×10^6 CAR+T, 3.0×10^6 CAR+T, 6.0×10^6 CAR+T
  Interventions: Drug: Human Derived anti-BCMA CAR-T Injection

INTERVENTIONS:
Drug: Human Derived anti-BCMA CAR-T Injection — Autologous genetically modified anti-BCMA CAR transduced T cells
  Other Names: BCMA CAR-T

SUMMARY:
This study is a single-arm, open-label, dose-escalation trial to explore the safety, tolerability and pharmacokinetic/pharmacodynamics characteristics of Human Derived anti-BCMA CAR-T Injection , and to preliminarily observe the efficacy of the trial drug in patients with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
Subjects withe relapsed/refractory multiple myeloma can participate if all eligibility criteria are met. Tests required to determine eligibility including disease assessments, a physical exam, Electrocardiograph, Computed tomography（CT）/Magnetic Resonance Imaging(MRI)/Positron Emission Tomography（PET）,liver/renal function tests, complete blood count with differential and complete metabolic profile and etc.. Subjects will receive precondtioning chemotherapy prior to the infusion of BCMA CAR- T cells. After the infusion, subjects will be followed for adverse events pharmacokinetic/pharmacodynamics characteristics, efficacy, of BCMA CAR-T cells. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:

Subjects must meet all of the following criteria to be enrolled:

* Subjects volunteer to participate in clinical trails, understand and inform the trials and sign informed consent form, be willing to complete all the trial procedures;
* 18 to 75 years old (including cut-off value), Male and female;
* Expected survival > 12 weeks;
* Previously diagnosed as multiple myeloma by IMWG updated criteria (2014);
* One of the following indicators is satisfied:

  1. Serum M protein: for immunoglobulin G (IgG) type , M protein≥ 10 g/L, or for immunoglobulin A (IgA) type , M protein > 5g/L, or for immunoglobulin D (IgD) type , M protein, IgD exceeds upper limit of normal range.
  2. Urine M protein ≥ 200 mg/24h;
  3. Serum free light chain ≥ 100 mg/L and Serum free light chain ratio is abnormal ;
* Patients with relapsed/refractory multiple myeloma. Relapsed is defined as: Patients have disease progression after at least three-line treatment regimens. Patients previously received at least 3 different mechanisms treatment regimens for multiple myeloma, including protease inhibitors and immunomodulators; Refractory is defined as: Patients who achieved minimal response(MR) or above was never achieved in previous treatment; MR or above was achieved in previous treatment, but disease progression occurred during subsequent treatment or within 60 days after the last treatment.
* ECOG score 0-2;
* Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. Creatinine clearance (estimated by Cockcroft Gault formula) ≥ 40 mL/min;
  2. Left ventricular ejection fraction >50%;
  3. Baseline peripheral oxygen saturation >95%;
  4. Total bilirubin ≤ 2×ULN; Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 × ULN;
* The venous access required for collection can be established and leukepheresis can be carriedaccording to the judgement of investigators.

Exclusion Criteria:

Any one of the following conditions cannot be selected as a subject：

* Accompanied by other uncontrolled malignancies;
* Subjects with positive Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) and peripheral blood Hepatitis B virus(HBV) DNA titer is ≥500IU/mL; hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; human immunodeficiency virus(HIV) antibody positive; syphilis primary screening antibody positive;
* Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure （New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease;
* Patients who are accounted to be not appropriate for this trail by investigator;
* Pregnant or lactating woman, and female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion;
* Received CAR-T treatment or other gene therapies before enrollment;
* Those who failed to sign informed consent form or comply with the research procedures; Unwilling or unable to comply with research requirements;
* Have had severe immediate hypersensitivity reactions to any drugs used in this research;
* Active or uncontrollable infection requiring systemic therapy within 14 days prior to enrollment;
* In the past two years, the terminal organ was damaged due to autoimmune diseases (such as Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus), or the systemic use of immunosuppressive or other systemic disease control drugs was required;
* Patients with symptoms of central nervous system.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-02-09 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity(DLT) | 28 days post infusion
  Safety Indicator

SECONDARY OUTCOMES:
Pharmacokinetics parameters - Maximum CAR level in blood and CAR level in bone marrow(Cmax) | 2 years post infusion
  Effectiveness Metrics
Pharmacokinetics parameters -Time to peak CAR level in blood (Tmax) | 2 years post infusion
  Effectiveness Metrics
Pharmacokinetics parameters - 28-day Area under the curve of the CAR level in blood(AUC0-28) | 2 years post infusion
  Effectiveness Metrics
Pharmacodynamics characteristics - Cytokines Concentrations,cytokines level in blood | 2 years post infusion
  Effectiveness Metrics
Pharmacodynamics characteristics -Clonal bone marrow plasma cells level | 2 years post infusion
  Effectiveness Metrics
Overall Response Rate (ORR) at 3 month post infusion | 3 month post infusion
  ORR defined as proportion of subjects who achieved Partial remission(PR) or better according to the International Myeloma Working Group response criteria (2016) (IMWG 2016) as determined by an Investigator assessment at 3 month post infusion.
Percentage of Subjects With Negative Minimal Residual Disease (MRD) | 2 years post infusion
  MRD negative rate is defined as the proportion of subjects who achieve MRD negative status
Duration of Subjects With Negative Minimal Residual Disease (MRD) | 2 years post infusion
  MRD duration will calculated among MRD negative responders fom the date of initial MRD negative to the date of first documented evidence of MRD positive, as defined in the IMWG criteria (2016).
Number of Subjects with Adverse Events | 2 years post infusion
  Adverse event is any untoward medical event that occurs in a subject administered an investigational drug.
Change from Baseline in Perform Status as Measured by Eastern Cooperative Oncology Group（ECOG）Score（0-4） | 2 years post infusion
  Eastern Cooperative Oncology Group（ECOG） Performance Status Score（0-4） will be assessed by the inverstigator at baseline and the respective time point, higher scores mean a worse performance status.
Change from Baseline in complete blood count with differential and blood biochemical examination | 2 years post infusion
  complete blood count with differential and blood biochemical examination will be assessed by the investigator at the respective time point.
Change from Baseline in Physical Exam | 2 years post infusion
  physical exam will be assessed by the inverstigator at the respective time poin.
Progression-free Survival (PFS) | 2 years post infusion
  PFS defined as time from date of initial infusion of CAR-T to date of first disease progression according to IMWG criteria (2016) , or death due to any cause, whichever occurs first.
Overall Survival (OS) | 2 years post infusion
  OS is measured from the date of the initial infusion of CAR-T to the date of the subject's death.
Duration of Response (DOR) | 2 years post infusion
  DOR will be calculated among responders (with a PR or better response) from the date of initial response (PR or better) to the date of first documented evidence of progressive disease, as defined in the IMWG criteria (2016).

OTHER OUTCOMES:
Distribution of CAR-T | 2 years post infusion
  CAR level in extramedullary lesions, pleural effusion, ascites, cerebrospinal fluid, etc, if appropriate.
Cytokines Concentrations | 2 years post infusion
  Cytokine levels in pleural effusion, ascites, cerebrospinal fluid, etc.if appropriate.
Different Expression Genes (DEGs) in Plasma Cells for Relapse Subjects as Measured by Single-cell Ribonucleic Acid (RNA) Sequencing. | 2 years post infusion
  Single-cell Ribonucleic Acid (RNA) Sequencing will be performed in relapsed subjects if appropriate. The different expression genes (DEGs) in plasma cells before and after relapse will be assessed by single-cell RNA sequencing, DEGs cutoff was adjusted p-value < 0.05 (Wilcoxon Rank Sum test) and the fold change >2.

CONTACTS AND LOCATIONS:
Overall Officials: Juan Du, Doctor, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China